CLINICAL TRIAL: NCT05454748
Title: Simultaneous Recording of Cognitive and Motor Functions After Stroke : Dissociation of Motor and Cognitive Deficits
Brief Title: Simultaneous Recording of Cognitive and Motor Functions After Stroke
Acronym: SACSO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Other Study IDs: D19-P043
Record Dates: First submitted 2022-06-27; First posted 2022-07-12 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2022-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy controls
- Stroke patients

SUMMARY:
Aim: To assess whether a cognitively demanding dual-task has greater impact on manual dexterity in chronic stroke patients than in healthy subjects.

Methods: A visuomotor force-tracking task, combining grip force and oculomotor recordings, will be applied in chronic stroke patients with mild-moderate hemiparesis without clinical cognitive impairments and in age-comparable healthy subjects. The dual-task includes avoiding visual distractors and mental addition of numbers. Dual-task effect is calculated as difference in force control accuracy (dual minus single-task) and as difference in saccade rate (addition of numbers minus visual distractors).

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* First symptomatic stroke more than 3 months ago
* Box and blocks test score < 52
* Mini Mental State Examination Test > 25

Exclusion Criteria:

* Psychiatric disease
* Risk of Pregnancy
* History of previous stroke
* Disability that may interfere with the performance of tasks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stroke patients group and Age comparable healthy controls group
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Saccade inhibition rate | Baseline measurement (one occasion)
  Cross sectional comparison of % of saccades performed towards visual distractors

CONTACTS AND LOCATIONS:
Locations (1):
- GHU Sainte Anne, Paris, France

REFERENCES:
- [Derived] Dziezuk E, Le Boterff Q, Van Ravestyn C, Mairesse S, Hamdoun S, Calvet D, Daghsen L, Carment L, Rosso C, Maier MA, Turc G, Mas JL, G Lindberg P. Divided attention and manual visuomotor control in stroke: a combined dual-task and eye movement study. J Neuroeng Rehabil. 2025 Oct 10;22(1):212. doi: 10.1186/s12984-025-01735-4. PMID 41074170